CLINICAL TRIAL: NCT00545740
Title: A Phase III, Randomised, Double-Blind, Dose-Response, Stratified, Placebo-Controlled Study Evaluating the Safety and Efficacy of SPD476 Versus Placebo Over 104 Weeks in the Prevention of Recurrence of Diverticulitis.
Brief Title: Prevention of Recurrence of Diverticulitis
Acronym: PREVENT1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPD476-313; 2007-004895-37 (EudraCT Number)
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SPD476 (1.2 g) (Experimental)
  Interventions: Drug: SPD476 (1.2g)
- SPD476 (2.4 g) (Experimental)
  Interventions: Drug: SPD476 (2.4 g)
- SPD476 (4.8 g) (Experimental)
  Interventions: Drug: SPD476 (4.8 g)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD476 (1.2g) — 1.2g SPD476 once daily (QD) orally
  Other Names: Lialda, MMX™ mesalazine
  Arms: SPD476 (1.2 g)
Drug: SPD476 (2.4 g) — 2.4g SPD476 QD orally
  Other Names: Lialda, MMX™ mesalazine
  Arms: SPD476 (2.4 g)
Drug: SPD476 (4.8 g) — 4.8g SPD476 QD orally
  Other Names: Lialda, MMX™ mesalazine
  Arms: SPD476 (4.8 g)
Drug: Placebo — QD orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether SPD476 is effective in reducing recurrence of diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females =>18yrs of age.
2. If female of childbearing potential (FOCP), has demonstrated a negative beta HCG (human chorionic gonadotropin) serum pregnancy test, and agrees to comply with any applicable contraceptive requirements of the protocol.
3. An episode of acute diverticulitis that resolved without colonic resection.
4. Confirmation of diverticulosis via endoscopic evaluation of the sigmoid colon with at least three diverticula noted.

Exclusion Criteria:

1. Previous colorectal surgery, including surgical intervention for diverticular disease (with the exception of haemorrhoidectomy, colonic removal of polyps, and appendectomy)
2. Active peptic ulcer disease
3. History of or current presence of inflammatory bowel disease (IBD)
4. Subjects with active irritable bowel syndrome (IBS) requiring ongoing medication
5. Allergy or hypersensitivity to aspirin or related compounds
6. Allergy to radiologic contrast agents
7. Use of another Investigational product within 30 days of Baseline
8. Use of antibiotic therapy within 4 weeks of Baseline
9. Within 14 days of Baseline, use of prebiotic, probiotic or 5-ASA medications, as well as drugs active at the 5HT-receptor or anti-spasmodic agents
10. Use of systemic or rectal steroids within 6 weeks of Baseline. Use of inhaled or nasal steroids is acceptable
11. Use of anti-inflammatory drugs, (NSIADs, COX-2 inhibitors) including aspirin (except for cardiac prophylaxis) and ibuprofen, on a regular and ongoing basis
12. History of alcohol or other substance abuse within the previous year
13. Active or recent history of endometriosis or dysmenorrhoea within 6 months prior to Baseline
14. Females who are lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2007-11-28 (Actual); Primary Completion 2012-03-05 (Actual); Study Completion 2012-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (121):
- United States (46):
  - Dedicated Clinical Research, Litchfield Park, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - GW Research, Chula Vista, California
  - Monterey Bay GI Research Institute, Inc, Monterey, California
  - Rancho Cucamonga C. Trials, Rancho Cucamonga, California
  - Clinical Trials Research, Roseville, California
  - Medical Associates Research, San Diego, California
  - Torrance Clinical Research, Torrance, California
  - Rocky Mountain Gastroenterology Associates, Thornton, Colorado
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - ZASA Clinical Research, Boynton Beach, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Compass Research, Orlando, Florida
  - Accord Clinic Research, LLC, Port Orange, Florida
  - Florida Medical Clinic/Tampa Clinical Trials, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Saint John's Research Institute, Anderson, Indiana
  - Digestive & Liver Disease Consultants, Clive, Iowa
  - New Orleans Research Institute, Metairie, Louisiana
  - Digestive Disease Associates, Baltimore, Maryland
  - Endoscopic Microsurgery Associates, PA, Towson, Maryland
  - Borgess Research Institute, Kalamazoo, Michigan
  - Jefferson City Medical Group, Jefferson City, Missouri
  - South Jersey Gastroenterology, P.A., Marlton, New Jersey
  - Howard Guss, DO, Ocean City, New Jersey
  - New Jersey Physicians, LLC, Passaic, New Jersey
  - Allied Gastrointestinal Associates, P.A., Voorhees Township, New Jersey
  - Regional Clinical Research, Endwell, New York
  - Long Island Clinical Research Associates, Great Neck, New York
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Research Associates of New York, New York, New York
  - Vital Research, Greensboro, North Carolina
  - Gastroenterology Specialists, Inc, Canton, Ohio
  - Memorial Research Center, Chattanooga, Tennessee
  - Gastroenterology Associates Clinical Research, Kingsport, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - Kelsey-Seybold Clinic, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Stone Oak Research Foundation, San Antonio, Texas
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Aurora Advanced Healthcare, Inc. - Clinical Research Center, Milwaukee, Wisconsin
- Argentina (7):
  - CIMEL, Lanús, Buenos Aires
  - Instituto Gamma, Rosario, Santa Fe Province
  - Hospital Bocalandro, Buenos Aires
  - Hospital Heroes de Malvinas, Buenos Aires
  - GEDYT, Buenos Aires
  - Sanatorio Guemes, Buenos Aires
  - Cibic S.A., Santa Fe
- Australia (8):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Ballarat Base Hospital, Ballarat, Victoria
  - St Vincent's Hospital (Melb) LTD, Melbourne, Victoria
  - Royal Adelaide Hospital, Adelaide
  - Royal Prince Albert Hospital, Camperdown
  - Frankston Private, Frankston
  - Bayside Gastroenterology, Frankston
  - Fremantle Hospital, Fremantle
- Colombia (6):
  - Ugasend S.A, Barranquilla
  - Clinica Colsinatas SA, Bogotá
  - FOQUS, Centro de Investigacion Clinica, Bogotá
  - Fundacion Clinica Abood Shaio, Bogotá
  - Hospital Universitario San Ignacio, Bogotá
  - Clinica Las Americas, Medellín
- France (10):
  - CHU de Strasbourg, Strasbourg, Alsace
  - CHU de Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - Hepato Gastro Enterology, Nantes, Brittany Region
  - Hopital Charles Nicolle, Rouen, Normandy
  - Hopital Beaujon, Clichy, Paris
  - Cabinet de Gastro-enterologie du Dr Alain Thevenin, Saint-Quentin, Picardie
  - Clinique Bouchard, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hopital I'Archet, Nice, Provence-Alpes-Côte d'Azur Region
  - Cabinet du Dr Olivier Delette, Lille
  - Dr Michel Regensberg, Paris
- India (10):
  - Baby Memorial Hospital, Calicut, Kerala
  - Lakeshore Hospital & Research Centre Ltd, Kochi, Kerala
  - Sree Gokulam Medical College and Research Foundation, Trivandrum, Kerala
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - S R Kalla Memorial Hospital, Jaipur, Rajasthan
  - Aceer, Chennai, Tamil Nadu
  - Institute of Postgraduate Medical Education and Research, Kolkata, West Bengal
  - Brahmin Mitra Mandal Society, Ahmedabad
  - Ruby Hall Clinic, Pune
  - Krishna Institute of Medical Sciences, Secunderabad
- Israel (12):
  - Emek Medical Center, Afula
  - Barzilai Medical Centre, Ashkelon
  - Soroka Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah Ein-Karem Medical Center, Jerusalem
  - Meir Medical Centre, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Ẕerifin
- New Zealand (6):
  - Shakespeare Specialist Group, Takapuna, Auckland
  - Auckland City Hospital, Auckland
  - CURT Medical Trials Trust Board, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Tauranga Hospital, Tauranga
- Spain (5):
  - Hospital Valle de Hebron, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital de Donostia, Donostia / San Sebastian
  - Hospital Son Dureta, Palma de Mallorca
  - Hospital General Universitario de Valencia, Valencia
- Sweden (6):
  - University Hospital/Eastern Hospital, Gothenburg
  - University Hospital Linköping, Linköping
  - VO Internmedicin, Stockholm
  - Karolinska University Hospital, Stockholm
  - Danderyd Hospital, Stockholm
  - Kirurgkliniken, Uppsala
- United Kingdom (5):
  - Norfolk/Norwich University Hospital, Norwich, East Anglia
  - St Mark's Hospital, Harrow, London
  - King's College Hospital, London
  - Chelsea & Westminster Hospital, London
  - Imperial College London, London

REFERENCES:
- [Derived] Raskin JB, Kamm MA, Jamal MM, Marquez J, Melzer E, Schoen RE, Szaloki T, Barrett K, Streck P. Mesalamine did not prevent recurrent diverticulitis in phase 3 controlled trials. Gastroenterology. 2014 Oct;147(4):793-802. doi: 10.1053/j.gastro.2014.07.004. Epub 2014 Jul 16. PMID 25038431

RESULTS

PARTICIPANT FLOW:
Groups:
- SPD476 (1.2 g): 1.2 g administered orally once daily
- SPD476 (2.4 g): 2.4 g administered orally once daily
- SPD476 (4.8 g): 4.8 g administered orally once daily
- Placebo: Placebo administered orally once daily
Period: Overall Study
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Started | 145 | 145 | 151 | 149
Completed | 70 | 62 | 55 | 78
Not Completed | 75 | 83 | 96 | 71
Not completed — Lack of Efficacy | 34 | 35 | 47 | 36
Not completed — Withdrawal by Subject | 17 | 15 | 16 | 18
Not completed — Adverse Event | 10 | 18 | 19 | 9
Not completed — Lost to Follow-up | 7 | 5 | 5 | 6
Not completed — Protocol Violation | 1 | 3 | 1 | 0
Not completed — Non-compliance | 0 | 2 | 1 | 0
Not completed — Moved | 2 | 0 | 1 | 0
Not completed — Diverticulitis attack | 0 | 0 | 1 | 1
Not completed — Suspected Diverticulitis Recurrence | 1 | 1 | 1 | 1
Not completed — Site closure | 1 | 0 | 0 | 0
Not completed — Missed visit | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 3 | 0
Not completed — Accepted only monthly telephone calls | 1 | 0 | 0 | 0
Not completed — Sponsor decision | 0 | 1 | 0 | 0
Not completed — Lack of time | 0 | 1 | 0 | 0
Not completed — Non-adherence to visits | 0 | 1 | 0 | 0
Not completed — Patient difficulties | 0 | 1 | 0 | 0
Not completed — Husband against study | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo | Total
Number analyzed (Participants) | 145 | 145 | 151 | 149 | 590
Age, Continuous [Mean (Standard Deviation); unit: years] — The Safety Population was used for this baseline measure. The Safety Population consists of subjects who were randomized and took at least 1 dose of investigational product. Out of the 590 subjects randomized, 7 were never dosed with investigational product. Therefore, 583 subjects are in the Safety Population.
  years | 55.1 (11.11) | 54.5 (11.96) | 54.5 (11.93) | 57.1 (10.42) | 55.3 (11.39)
Age, Customized [Count of Participants; unit: Participants] — The Safety Population was used for this baseline measure. The Safety Population consists of subjects who were randomized and took at least 1 dose of investigational product. Out of the 590 subjects randomized, 7 were never dosed with investigational product. Therefore, 583 subjects are in the Safety Population.
  Participants
    18 to <35 years | 3 | 11 | 8 | 3 | 25
    35 to <45 years | 20 | 17 | 26 | 14 | 77
    45 to <55 years | 49 | 39 | 36 | 37 | 161
    55 to <65 years | 43 | 46 | 51 | 62 | 202
    >= 65 years | 28 | 30 | 29 | 31 | 118
Sex/Gender, Customized [Count of Participants; unit: Participants] — The Safety Population was used for this baseline measure. The Safety Population consists of subjects who were randomized and took at least 1 dose of investigational product. Out of the 590 subjects randomized, 7 were never dosed with investigational product. Therefore, 583 subjects are in the Safety Population.
  Participants
    Female | 64 | 69 | 71 | 71 | 275
    Male | 79 | 74 | 79 | 76 | 308
Region of Enrollment [Count of Participants; unit: Participants] — This baseline measure consists of all randomized subjects (n = 590).
  Participants
    Argentina | 5 | 3 | 4 | 3 | 15
    Australia | 3 | 5 | 6 | 5 | 19
    Colombia | 19 | 18 | 18 | 19 | 74
    France | 5 | 6 | 6 | 6 | 23
    India | 4 | 2 | 3 | 4 | 13
    Israel | 24 | 24 | 23 | 24 | 95
    New Zealand | 3 | 4 | 4 | 4 | 15
    Spain | 1 | 1 | 4 | 2 | 8
    Sweden | 9 | 9 | 11 | 9 | 38
    United Kingdom | 3 | 3 | 3 | 4 | 13
    United States | 69 | 70 | 69 | 69 | 277

OUTCOME MEASURES:

1. Secondary Outcome: Percent of Subjects Who Were CT-Recurrence Free of Diverticulitis
Description: CT-recurrence of diverticulitis is defined as: a positive spiral CT scan for diverticulitis showing, at a minimum, fat stranding with or without bowel wall thickening >5 mm or surgical intervention for diverticular disease. Withdrawals considered as CT-recurrences.
Time Frame: Up to 104 weeks
Population: Full Analysis Set (FAS) consists of all subjects who were randomized and took at least 1 dose of investigational product.
Measure: Number; unit: percentage of subjects
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 143 | 143 | 150 | 147
percentage of subjects | 61.5 | 62.2 | 52.7 | 63.9
Statistical Analysis 1: Comparison: SPD476 (4.8 g) vs Placebo; Test type: Superiority or Other; p = 0.063, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SPD476 (2.4 g) vs Placebo; Test type: Superiority or Other; p = 0.736, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SPD476 (1.2 g) vs Placebo; Test type: Superiority or Other; p = 0.780, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of CT Scans Performed Within 7 Days of Suspected Recurrence of Diverticulitis That Were Positive
Description: A positive CT scan was defined as a CT scan that showed bowel wall thickening (>5 mm) and/or fat stranding as read by the central reader.
Time Frame: Up to 104 weeks
Population: Suspected Recurrence of Diverticulitis consists of subjects in the Full Analysis Set who had a CT scan performed. Since subjects may have had more than one suspected recurrence, counts are of the number of CT scans, not the number of subjects.
Measure: Number; unit: Number of CT scans
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 52 | 49 | 55 | 46
Number of CT scans
  Positive | 37 | 39 | 55 | 38
  Presence of abdominal pain | 30 | 39 | 54 | 37
  15% increase in WBC from baseline | 17 | 24 | 28 | 24
  Presence in abdominal pain + 15% increase in WBC | 17 | 24 | 28 | 23

3. Primary Outcome: Percent of Subjects Without Recurrence of Diverticulitis
Description: Recurrence of diverticulitis is defined as the presence of each and all of the following 3 items: 1) abdominal pain, 2) a 15% increase in white blood cell count from baseline, 3) bowel wall thickening (>5 mm) and/or fat stranding as evidenced by spiral computerized axial tomography (CT) scan; OR surgical intervention for diverticular disease. Withdrawals are considered as recurrences.
Time Frame: Up to 104 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 143 | 143 | 150 | 147
percentage of subjects | 62.2 | 62.9 | 52.7 | 64.6
Statistical Analysis 1: Comparison: SPD476 (4.8 g) vs Placebo; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SPD476 (2.4 g) vs Placebo; Test type: Superiority or Other; p = 0.741, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SPD476 (1.2 g) vs Placebo; Test type: Superiority or Other; p = 0.780, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of CT Scans Performed Within 7 Days of Suspected Recurrence of Diverticulitis That Were Negative
Description: A negative CT scan was defined as a CT scan that did not show bowel wall thickening (>5 mm) and/or fat stranding as read by the central reader.
Time Frame: Up to 104 weeks
Population: as for outcome 2
Measure: Number; unit: Number of CT scans
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 52 | 49 | 55 | 46
Number of CT scans
  Negative | 19 | 10 | 5 | 10
  Presence of abdominal pain | 19 | 8 | 5 | 7
  15% increase in WBC from baseline | 5 | 2 | 2 | 1
  Presence in abdominal pain + 15% increase in WBC | 5 | 2 | 2 | 1

5. Secondary Outcome: Number of CT Scans Performed More Than 7 Days From Suspected Recurrence of Diverticulitis That Were Positive
Description: as for outcome 2
Time Frame: Up to 104 weeks
Population: as for outcome 2
Measure: Number; unit: Number of CT scans
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 52 | 49 | 55 | 46
Number of CT scans
  Positive | 0 | 0 | 1 | 1
  Presence of abdominal pain | 0 | 0 | 1 | 1
  15% increase in WBC from baseline | 0 | 0 | 0 | 0
  Presence of abdominal pain + 15% increase in WBC | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of CT Scans Performed More Than 7 Days From Suspected Recurrence of Diverticulitis That Were Negative
Description: as for outcome 4
Time Frame: Up to 104 weeks
Population: as for outcome 2
Measure: Number; unit: Number of CT scans
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 52 | 49 | 55 | 46
Number of CT scans
  Negative | 0 | 3 | 2 | 3
  Presence of abdominal pain | 0 | 2 | 2 | 3
  15% increase in WBC from baseline | 0 | 1 | 0 | 1
  Presence of abdominal pain + 15% increase in WBC | 0 | 0 | 0 | 1

7. Secondary Outcome: Percent of Subjects Requiring Surgery for Diverticulitis
Time Frame: Up to 104 weeks
Population: Full Analysis Set consists of all subjects who were randomized and took at least 1 dose of investigational product.
Measure: Number; unit: percentage of subjects
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 143 | 143 | 150 | 147
percentage of subjects | 2.8 | 2.8 | 3.3 | 2.0

ADVERSE EVENTS:
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Serious Adverse Events (participants affected / at risk) | 16/143 | 15/143 | 18/150 | 16/147
Other Adverse Events (participants affected / at risk) | 109/143 | 106/143 | 101/150 | 112/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPD476 (1.2 g) (N=143) | SPD476 (2.4 g) (N=143) | SPD476 (4.8 g) (N=150) | Placebo (N=147)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 1 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocarcial infarction (Cardiac disorders) | 1 | 0 | 0 | 2
Coronary artery insufficiency (Cardiac disorders) | 1 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peritoneal hematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Near drowning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ischemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Movement disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral ischemia (Nervous system disorders) | 0 | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 0 | 1 | 0
Bipolar II disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD476 (1.2 g) (N=143) | SPD476 (2.4 g) (N=143) | SPD476 (4.8 g) (N=150) | Placebo (N=147)
Abdominal pain (Gastrointestinal disorders) | 17 | 16 | 18 | 16
Diarrhea (Gastrointestinal disorders) | 13 | 12 | 12 | 12
Nausea (General disorders) | 10 | 1 | 6 | 5
Flatulence (Gastrointestinal disorders) | 9 | 5 | 3 | 4
Constpation (Gastrointestinal disorders) | 7 | 3 | 5 | 8
Urinary tract infection (Infections and infestations) | 14 | 12 | 8 | 17
Nasopharyngitis (Infections and infestations) | 6 | 15 | 7 | 13
Upper respiratory tract infection (Infections and infestations) | 9 | 3 | 10 | 14
Sinusitis (Infections and infestations) | 9 | 7 | 5 | 8
Influenza (Infections and infestations) | 5 | 11 | 4 | 3
Bronchitis (Infections and infestations) | 7 | 8 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5 | 8 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 4 | 13
Headache (Nervous system disorders) | 13 | 6 | 14 | 10
Hypertension (Vascular disorders) | 5 | 8 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.